CLINICAL TRIAL: NCT06515431
Title: Myocardial Injury After Radical Nephrectomy
Acronym: MANE
Status: Withdrawn | Type: Observational
Why Stopped: not feasible
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH22687
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic nephrectomy
- Robotic nephrectomy

SUMMARY:
Kidney removal for cancer (nephrectomy) is a major operation. People can develop heart complications during or after surgery, especially if they are older or already have heart disease. One form of heart damage is called myocardial injury (MINS). This can be detected with a simple and easily available blood test. Unlike a heart attack, MINS doesn't cause changes in the electrical tracing of the heart (ECG) and it typically doesn't cause symptoms like pain. However, it can lead to heart problems and a stroke after surgery. We do not know how many people having a nephrectomy develop MINS. It is important to know if people are at high risk of MINS to help decide future treatment.

There are a few different ways of carrying out nephrectomy surgery. These can be traditional open surgery, keyhole surgery or robotic surgery. We know that MINS is more likely if there has been a lot of bleeding during the operation, but other factors are also important. Therefore, it's important to monitor the relationship between blood loss, rates of MINS and method of surgery.

We aim to recruit 120 participants undergoing nephrectomy to see how many develop MINS and to compare blood loss between different ways of surgery. Patients will be asked to consent to have blood tests on the day of and the day after surgery. This test will be added to routine hospital blood tests (and so no extra samples are needed). These results will show how many patients are diagnosed with MINS after nephrectomy. Around 90 days after the surgery, their quality of life and any further heart or breathing problems will also be recorded.

We hope to identify the rates of and risk factors for MINS, so future patients can be spared this complication of surgery.

DETAILED DESCRIPTION:
Patients undergoing nephrectomy have a greater risk of cardiac events requiring admission compared to the general population. For example, registry data report 21% of patients over 65 undergoing nephrectomy have at least one cardiovascular event after surgery. Myocardial injury after non-cardiac surgery (MINS) is a condition which is associated with increased mortality and a higher rate of major adverse cardiac events (MACE), in both the immediate perioperative period and within 1-year post-surgery. Diagnosis is via the presence of elevated troponin levels in the first 3 days post-surgery, in the absence of ischaemic symptoms and ECG changes.

The occurrence of MINS following nephrectomy for renal cell carcinoma has not yet been explored. Risk factors for MINS include increasing age and post-operative acute kidney injury. Results from the British Association of Urological Surgeons (BAUS) Nephrectomy audit demonstrate that most patients undergoing nephrectomy are over 60 and that increasing age is associated with lower eGFR pre-operatively. The accepted further reduction in post-operative GFR with nephrectomy makes these patients at high risk of MINS.

The BAUS Nephrectomy audit also demonstrates that elderly patients undergoing nephrectomy are likely to be anaemic preoperatively. In at-risk patients, any intraoperative haemodynamic instability may progress to myocardial injury and cardiac related complications due to a change in myocardial oxygen demand.

Most radical nephrectomies are now performed using robotic or laparoscopic approaches. Current evidence from retrospective studies and a small prospective study suggests that there is no difference in perioperative nor oncological outcomes between laparoscopic and robotic radical nephrectomy, including blood loss. However, no studies to date have looked at MINS and large-scale prospective studies comparing the haemodynamic effects of laparoscopic vs robotic nephrectomy are needed.

Understanding the spectrum of MINS and its potential impact on patients undergoing nephrectomy is pivotal. This could lead to better patient selection and stratified care to improve outcomes. Advances in systemic therapy for metastatic disease mean nephrectomy may become more prevalent in persons on multiple therapies. As patients undergoing nephrectomy are at high risk of MINS, it is vital to have a greater understanding of this potential complication. This aligns with the James Lind Alliance Priority Setting Partnership in perioperative care which highlights the importance of research into post-operative complications. Furthermore, this group also underlines the importance of adequate preoperative discussions with patients, which would include the risk of postoperative complications such as MINS.

Eligible patients who have consented to the study will have their troponin levels measured on the day of the surgery and at day 1 post-op to diagnose MINS. A baseline quality of life assessment will also be made by asking patients to complete an EQ-5D-5L questionnaire. Any blood transfusions during the admission period will also be recorded. At day 90 post-op, the occurrence of MACE events and days out of hospital (DAOH90) will be checked, and the patient will be contacted to complete the quality-of-life questionnaire again.

Baseline assessments:

The following demographic information will be prospectively collected by reviewing the patient's medical notes:

* Age, sex, and ethnicity
* Previous history of ischaemic heart disease, congestive cardiac failure, cerebrovascular disease (stroke or TIA), diabetes
* Tumour characteristics (radiological T stage, laterality)

Pre-op renal function and baseline troponin will be measured on the day of surgery.

Primary outcome measure:

The primary outcome measure is the proportion of patients undergoing laparoscopic or robotic radical nephrectomy with evidence of myocardial injury (MINS). This will be defined as a raised troponin level >99th percentile upper reference limit on any sample taken within 72 hours following the operation.

Patients will have troponin levels measured on the morning of surgery and at day 1 post-op. If applicable, this can be retrieved as an 'add on' test on routine samples, without the requirement for an additional "blood draw" to avoid extra burden to patients.

Sites will be expected to manage patients post-operatively as per Trust guidelines - this may or may not include troponin monitoring. The European Society for Cardiology advocates testing of troponins but does not make treatment recommendations. If troponin monitoring is not part of usual care, the troponin samples will not be available to the clinical team to avoid any inadvertent additional investigations which may add to patient burden. Instead, we would arrange the troponin results to be processed after surgery.

However, the clinical team can request troponin tests for clinical information, for example in the assessment of chest pain. In this situation, the troponin sample would be processed immediately and be available for the clinical team to view. The clinical team will be expected to follow local guidelines regarding the clinical management. If the clinical team requests a troponin level for clinical assessment, we will also note this in the research record.

Secondary outcome measures:

Perioperative assessments:

● Any blood transfusions during the intraoperative and/or postoperative period will be recorded. This will allow assessment of potential cardiovascular instability compared between the groups (laparoscopic vs robot-assisted) and how this translates to rates of MINS and MACE post-op.

90 days (+/- 7 days) post-procedure:

Patients will be contacted by the research team via telephone to assess the following:

* The occurrence of any major adverse cardiovascular event (myocardial infarction, stroke, arrhythmia, cardiac arrest, and cardiac related death) during admission will be recorded. This will be obtained as part of patient follow up at 90 days post-op.
* Days out of hospital at 90 days (DAOH90). This will be recorded following discussion with the patient and review of local hospital data
* Impact on quality of life will be assessed using the EQ-5D-5L via a telephone interview by the research team.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (aged 18 and above)
* Undergoing a radical nephrectomy (either laparoscopic or robotic) for suspected renal cancer
* Stage <T3a
* Can provide informed consent

Exclusion Criteria

* Patients under 18
* Undergoing partial nephrectomy
* Undergoing radical nephrectomy not for suspected renal cancer
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery waiting lists will be screened by members of the research team at Sheffield Teaching Hospitals to identify patients that will be undergoing a radical nephrectomy for suspected renal cancer. The surgical approach will already have been decided before the study is introduced. Those eligible will be contacted via phone to discuss the study further.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients undergoing radical nephrectomy with evidence of myocardial injury (MINS) | 72 hours post surgery
  This will be defined as a raised troponin level >99th percentile upper reference limit on any sample taken within 72 hours following the operation.

SECONDARY OUTCOMES:
Occurrence of intraoperative and post-operative blood transfusion | 72 hours post surgery
Number of days out of hospital | 90 days post surgery
Rate of major adverse cardiac events (MACE) | 90 days post surgery
  MACE events are defined as (myocardial infarction, stroke, arrhythmia, cardiac arrest, and cardiac related death
Impact on quality of life, assessed by EQ-5D-5L questionnaire completed by patients | 90 days post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No